CLINICAL TRIAL: NCT00458705
Title: Bortezomib + Pegylated Liposomal Doxorubicin (Doxil) + Dexamethasone Followed by Thalidomide + Dexamethasone or Bortezomib + Thalidomide + Dexamethasone for Patients With Symptomatic Untreated High-Risk or Primary Resistant Multiple Myeloma
Brief Title: Bortezomib, Doxorubicin Hydrochloride Liposome, and Dexamethasone Followed by Thalidomide and Dexamethasone With or Without Bortezomib in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-067; P30CA008748 (NIH); MSKCC-06067
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Results first posted 2016-01-22 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2015-12

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Bortezomib; Dexamethasone; Thalidomide

ARMS (1):
- Combination therapy (Experimental): Combination therapy with bortezomib, pegylated liposomal doxorubicin and dexamethasone (BDD) followed by either thalidomide and dexamethasone (TD) or bortezomib, thalidomide and dexamethasone in patients with symptomatic untreated high-risk or primary resistant multiple myeloma. Three cycles of BDD will be administered. Patients who respond after three cycles will receive two cycles of TD. Patients with stable or progressive disease after three cycles of BDD receive two cycles of bortezomib, thalidomide and dexamethasone. If at any point during the study a patient achieves a complete response (CR), the patient will be given the option to discontinue treatment on-study.
  Interventions: Drug: bortezomib; Drug: dexamethasone; Drug: pegylated liposomal doxorubicin hydrochloride; Drug: thalidomide

INTERVENTIONS:
Drug: bortezomib
Drug: dexamethasone
Drug: pegylated liposomal doxorubicin hydrochloride
Drug: thalidomide

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as doxorubicin hydrochloride liposome and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or stopping them from dividing. Thalidomide may stop the growth of cancer cells by blocking blood flow to the cancer. Giving bortezomib together with doxorubicin hydrochloride liposome and dexamethasone followed by thalidomide, dexamethasone, and bortezomib may kill more cancer cells.

PURPOSE: This phase II trial is studying the side effects and how well giving bortezomib together with doxorubicin hydrochloride liposome and dexamethasone followed by thalidomide and dexamethasone with or without bortezomib works in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy and safety of bortezomib, pegylated doxorubicin hydrochloride liposome, and dexamethasone followed by thalidomide and dexamethasone with or without bortezomib in patients with symptomatic high-risk or primary resistant multiple myeloma.

OUTLINE: Patients receive BDD comprising bortezomib IV on days 1, 4, 8, and 11; pegylated doxorubicin hydrochloride liposome IV over 60-90 minutes on day 4; and oral dexamethasone on day 1, 2, 4, 5, 8, 9, 11, and 12. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.

Patients achieving response to BDD receive oral thalidomide on days 1-28 and oral dexamethasone on days 1-4, 9-12, and 17-20. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity.

Patients experiencing stable or progressive disease on BDD receive oral thalidomide on days 1-28; oral dexamethasone on days 1, 2, 4, 5, 8, 9, 11, 12, and 17-21; and bortezomib IV on days 1, 4, 8, and 11. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically and serologically confirmed multiple myeloma meeting one of the following criteria:

  * High-risk myeloma, defined as symptomatic International Staging System (ISS) stage 2 or 3 multiple myeloma
  * Soft-tissue involvement with myeloma in the form of a soft-tissue plasmacytoma
  * Extension of a plasmacytoma into soft tissues
  * Primary resistant myeloma, defined as unchanged or progressive myeloma despite two courses of standard treatment
* No ISS stage 1 multiple myeloma without soft-tissue involvement
* No smoldering myeloma

PATIENT CHARACTERISTICS:

* ECOG performance status 0-3
* Life expectancy > 16 weeks
* Absolute granulocyte count ≥ 1,500/mm³ (unless low granulocyte counts are due to multiple myeloma)
* Platelet count ≥ 100,000/mm³ (unless low platelet counts are due to multiple myeloma)
* Bilirubin ≤ 2.0 mg/dL
* AST and ALT < 3 times upper limit of normal (ULN)
* Alkaline phosphatase < 3 times ULN
* LVEF ≥ 50% by MUGA or ECHO
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception 4 months prior to, during, and for 4 weeks after completion of study treatment
* No active thromboembolic disease on anticoagulation
* No active angina or myocardial infarction within the past 6 months
* No pre-existing neuropathy or sensory or neuropathic pain ≥ grade 2
* No concurrent active malignancy other than nonmelanoma skin cancer or carcinoma in situ of the cervix

  * Prior malignancies that have not required antitumor treatment within the past 24 months allowed
  * Patients with a history of stage I or II (T1a/b) prostate cancer (detected incidentally at transurethral resection of prostate [TURP] and comprising < 5% of resected tissue) allowed if the prostate-specific antigen has remained normal since TURP
* No known HIV positivity or AIDS-related illness
* No other medical condition or reason that, in the opinion of the investigator, would preclude study compliance
* No history of hypersensitivity reactions attributed to a conventional formulation of doxorubicin hydrochloride or to components of pegylated doxorubicin hydrochloride liposome, bortezomib, boron, or mannitol

PRIOR CONCURRENT THERAPY:

* Prior radiotherapy allowed
* No more than 2 courses of prior initial chemotherapy for multiple myeloma
* No prior bortezomib
* No prior high-dose steroids (not including taper) for more than 1 month in duration for emergent indications, such as hypercalcemia or life-threatening lesions (e.g., spinal cord compromise) (in high-risk patients)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Landau, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Landau H, Pandit-Taskar N, Hassoun H, Cohen A, Lesokhin A, Lendvai N, Drullinsky P, Schulman P, Jhanwar S, Hoover E, Bello C, Riedel E, Nimer SD, Comenzo RL. Bortezomib, liposomal doxorubicin and dexamethasone followed by thalidomide and dexamethasone is an effective treatment for patients with newly diagnosed multiple myeloma with Internatinal Staging System stage II or III, or extramedullary disease. Leuk Lymphoma. 2012 Feb;53(2):275-81. doi: 10.3109/10428194.2011.606943. Epub 2011 Sep 23. PMID 21824051

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combination Therapy
Started | 45
Completed | 40
Not Completed | 5
Not completed — Adverse Event | 4
Not completed — Not Treated | 1

BASELINE CHARACTERISTICS:
Arm/Group | Combination Therapy
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 30
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Disease Response
Description: The response of myeloma to BDDTD will be assessed by standard electrophoretic and immunofixation tests of blood and urine for a monoclonal protein (M protein), and bone marrow aspirate and biopsy. These tests will be performed at enrollment and at the conclusion of therapy.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Combination Therapy
Number analyzed (Participants) | 40
participants
  Complete Response | 10
  Near Complete Response | 8
  Partial Response | 10
  Stable Disease | 2
  Progression of Disease | 3
  Very Good Partial Response | 7

ADVERSE EVENTS:
Arm/Group | Combination Therapy
Serious Adverse Events (participants affected / at risk) | 22/45
Other Adverse Events (participants affected / at risk) | 23/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy (N=45)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Creatinine increased (Investigations) | 1 (1)
Death not assoc w CTCAE term- Multi-organ failure (General disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Fever (General disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hepatobiliary disorders -other, specify (Hepatobiliary disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Infection (Infections and infestations) | 3 (3)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Lymphocyte count decrease (Investigations) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Neuralgia (Nervous system disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders-other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal and urinary disorders -other, specify, Renal failure (Renal and urinary disorders) | 5 (5)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 6 (7)
Urinary retention (Renal and urinary disorders) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy (N=45)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Neuralgia (Nervous system disorders) | 4 (6)
Renal and urinary disorders -other, specify-Renal failure (Renal and urinary disorders) | 4 (4)
Thrombosis/thrombus/embolism (Vascular disorders) | 8 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes